CLINICAL TRIAL: NCT05395897
Title: ORiginal meThodology for Assessing the Impact of the Coronavirus Health Crisis on Psychotropic Drug Use
Acronym: TORNADO
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0409
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Psychotropic Drugs
Keywords: Psychotropic drugs, SARS-CoV-2, health impact assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New users: Users without any reimbursement for psychotropic drugs before the beginning of the coronavirus crisis.
- Actual or former users: Users without at least one reimbursement for psychotropic drugs before the beginning of the coronavirus crisis.

SUMMARY:
The health crisis linked to the coronavirus has had a significant impact on the mental health. The question of the repercussion of this crisis on the consumption of psychotropic drugs is crucial. It is all the more true in France, which was already among the countries with the highest consumption of psychotropic drugs before the crisis. Indeed, an increase in the number of reimbursements for anxiolytic, hypnotic and antidepressant drugs has been highlighted in the context of the health crisis, using data from the health insurance database.

To enhance the understanding about the impacts of the health crisis on the use of psychotropic drugs, it is essential to characterize the evolution of the use at the individual level.

The main objective is to assess the impact of the coronavirus-related health crisis on the consumption of psychotropic drugs by studying the trajectories of reimbursements.

The secondary objective of the project is to evaluate the evolution of problematic consumption of psychotropic drugs in the context of the health crisis.

DETAILED DESCRIPTION:
The project will allow studying the evolution of the use of psychotropics since the coronavirus-related health crisis according to the temporality of consumption (succession and/or concomitance of consumption) or their persistence over time.

This project has two major aims:

* Pharmacosurveillance: evaluation of the impact of psychotropic drug consumption in the context of the health crisis related to the coronavirus. The consumption of psychotropic drugs is a public health issue in France and concerns the entire general population. Even before the crisis, France was one of the countries in the world where the consumption of psychotropic drugs was the highest.
* Scientific: use of an innovative methodology for assessing the impact of pharmaco-epidemiology (trajectories based on reimbursement data).

ELIGIBILITY:
Inclusion Criteria:

* Subjects identified in the French National Healthcare Data System (SNDS) in 2018, 2019, 2020 and 2021 at national level, alive on 01/01/2018, age ≥ 16 years on 01/01/2020.

Exclusion Criteria:

* Institutionalization at least one day in a residential facility for dependent elderly people with an internal pharmacy in 2018, 2019, 2020 or 2021.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A 10% random sample of the subjects identified in the SNDS, weighted on the region of residence.
Sampling Method: Probability Sample
Enrollment: 2772093 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Trajectories of healthcare consumption (psychotropic drugs, consultations, hospitalizations) | 2020-2021
  Trajectories will be defined as the succession of healthcare events. Multidimensional trajectories will be constructed taking into account the timing and concomitance of reimbursements

SECONDARY OUTCOMES:
Problematic use of psychotropic drugs | 2018-2021
  The evolution of indicators of problematic use for psychotropic drugs will be studied: doctor shopping, pharmacy shopping, overconsumption

CONTACTS AND LOCATIONS:
Overall Officials: Caroline VIGNEAU, Professor, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes university hospital, Nantes, Loire-atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided